CLINICAL TRIAL: NCT06029322
Title: A Randomized Controlled Trial Comparing Collagen Matrix to Collagen Membrane as Socket Seal in Alveolar Ridge Preservation
Brief Title: A Comparative Clinical Study Between a Collagen Matrix and Collagen Membrane as Wound Protection During Ridge Preservation ARP
Acronym: ARP
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: ONZ-2023-0516
Record Dates: First submitted 2023-08-31; First posted 2023-09-08 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Oral Soft Tissue Conditions
Keywords: collagen matrix; collagen membrane; alveolar ridge preservation (ARP); CBCT analysis; Volumetric analysis; peri-implant health; oral implant

STUDY DESIGN:
Intervention Model Description: Split-mouth design, intra-subject RCT Patients receive both treatments: collagen matrix and collagen membranes
Who Masked: Investigator, Outcomes Assessor
Masking Description: It concerns a surgical intervention. Hence, the treating surgeon and patient cannot be masked. The investigators and outcome assessors are masked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Collagen membrane (Active Comparator): BioGide Compressed® 13x25 mm, Geistlich Pharma AG, Wolhusen, Switzerland
  Interventions: Procedure: Socket seal after alveolar ridge preservation
- collagen matrix (Experimental): Mucograft Seal®, Geistlich Pharma AG, Wolhusen, Switzerland
  Interventions: Procedure: Socket seal after alveolar ridge preservation

INTERVENTIONS:
Procedure: Socket seal after alveolar ridge preservation — Socket seal is performed after ARP. Using a collagen matrix or membrane the socket is sealed, at the control (membrane) site a small pouch is made at the buccal and lingual aspect. Monofilament sutures are used to secure the respective material in place.

SUMMARY:
Patients in need of extraction of two teeth in combination with alveolar ridge preservation will be invited to participate in intra-subject RCT on ARP. Prior to surgery, a small-field low-dose CBCT is taken.

18 patients will be included, each contributing 1 surgical site to each treatment arm.

Since this study is a intra-subject RCT randomization of the surgical site will be performed just after ARP by a coin flip. Randomization is concealed for the evaluating examiner and statistician.

After ARP the collagen matrix or collagen membrane is used to seal the coronal aspect of the extraction socket.

Soft tissue thickness in centre of the site will be determined using CBCT. Secondary outcomes include: Wound dimensions, socket wound healing score, changes in bone and soft tissue dimensions and changes in buccal soft tissue profile

DETAILED DESCRIPTION:
The primary study objective is to compare soft tissue thickness in the centre of the site between collagen matrix and collagen membrane at 4 months following ARP.

Secondary study outcomes relate to the same comparison and include the following variables: wound reduction after 7 days and 21 days, socket wound healing score after 7 days, 21 days and 4 months, changes in bone and soft tissue dimensions including soft tissue profile between pre-op and 4 months.

Patients will be included in an intra-subject RCT on ARP following screening and written consent at the Department of Periodontology and Oral Implantology of the University Hospital in Ghent.

A sample size calculation was performed in SPSS Statistics 28 (IBM, New York, USA) using the paired samples t-test. The calculation was based on finding a mean difference of 0.5 mm in the final soft tissue thickness between test and control sites with a standard deviation of 0.6 mm (Eeckhout et al., 2022). With alpha set at 0.05 and a power of 0.08, the sample size calculation indicated 14 patients to be included. To compensate for possible dropouts, this number was increased to 18 patients.

Randomization, allocation concealment and blinding Since this is an intra-subject RCT, every patient receives the test treatment as well as the control treatment. A coin flip will determine which site in each patient is treated with the collagen matrix (test site) and which one with the collagen membrane (control site). Group allocation will be determined just after ARP and remains concealed for the evaluating examiner and statistician to allow for unbiased registrations and analyses, respectively.

Treatment procedures and postoperative care Patients will be instructed to take systemic antibiotics (amoxicilline 2g) and anti-inflammatory medication (ibuprofen 600 mg) 1 h pre-operatively. Just prior to the treatment, patients rinse with a 0.12% chlorhexidine solution (Perio-aid® Intensive Care, Dent-Aid Benelux, Houten, The Netherlands) and local anesthesia (Septanest special®, noradrenaline 1/100000; Septodont, Saint Maur des Fossés, France) will be administered.

Teeth are preferably extracted without flap elevation. When deemed necessary by the clinician, papillary incisions can be made for minimal reflection, which enables to place elevators without damaging soft tissues. Buccal soft tissues must never be raised. Following wound debridement and rinsing, the amount of missing bone is measured with a periodontal probe to the nearest 0.5 mm. Missing buccal bone is defined as the vertical distance between the buccal bone crest and the midfacial soft tissue margin minus 3 mm. Then, both alveolar sockets are filled with collagen-enriched deproteinized bovine bone mineral (C-DBBM, Bio-Oss Collagen® 100 mg or 250 mg, Geistlich Pharma AG, Wolhusen, Switzerland) up to the level of the lingual bone crest. The same procedure is performed for intact and non-intact alveoli. Thereupon, a coin will be flipped to determine the assignment for either one of two treatment modalities to each site:

* Test site: collagen matrix (Mucograft Seal®, Geistlich Pharma AG, Wolhusen, Switzerland)
* Control site: collagen membrane (BioGide Compressed® 13x25 mm, Geistlich Pharma AG, Wolhusen, Switzerland) At the control site a small pouch is made at the buccal and lingual aspect in order to place the membrane. The socket seal material is sutured with at least 4 single sutures (Seralon 6/0, Serag Weissner, Naila, Germany) to protect the underlying C-DBBM. Care is taken to ensure perfect approximation between the wound margins and the socket seal material.

Systemic antibiotics (amoxicilline 2g) will be continued for 4 days and anti-inflammatory medication (ibuprofen 600 mg) is taken as deemed necessary by the patient. Patients rinse with a 0.12% chlorhexidine solution twice daily for 1 week. Then, sutures are removed.

Primary outcome: soft tissue thickness in the centre of the site Soft tissue thickness in the centre of the site will be assessed using the method of Seyssens et al. (2019). A small-field low-dose CBCT image is taken at T0 (immediately postop) and T3 (4 months). All CBCT images will be obtained using a ProMax 3D Max device (Planmeca, Helsinki, Finland) with the same standardized settings (90 kV, 6.3 mA, 9 seconds, voxel size 200 μm) with a same field of view 50 × 80 mm for each patient. Lip retractors are used to clearly visualize the external soft tissue profile and patients will be instructed to fold the tongue backwards for the same reason. Using specialized software (Invivo6, Osteoid Inc., Santa Clara, California, United States), both CBCT images are superimposed. First, a reference line is drawn on the postoperative CBCT (T0) at the level of the long axis of the extracted tooth. Then, the software switch to the superimposed CBCT (T3) while keeping this reference line. Soft tissue thickness in the centre of the site will be measured on the reference line as the vertical distance between the alveolar proces and the soft tissue outline.

Bucco-lingual and mesio-distal wound dimensions These are registered with a periodontal probe to the nearest 0.5 mm at T0 (immediately postop), T1 (1 week) and T2 (3 weeks).

Socket Wound Healing Score (SWHS) SWHS (Afat et al., 2019) is assessed at T1 (1 week), T2 (3 weeks) and T3 (4 months). SWHS is used to evaluate wound dehiscence, epithelialization, quality of granulation tissue filling the post-extraction socket, and depth between early granulation tissue and wound margin. SWHS is assessed on the basis of occlusal clinical pictures and results in the following scores: 0 = Wound covered with keratinized gingiva, pink tissue color, no bleeding, continuous with healthy tissue; 1 = Socket filled with organized granulation tissue, no bleeding, collapsed to a depth of 0 - 2 mm from the buccal gingival margin; 2 = Socket filled with organized granulation tissue, ¼ to ½ of the wound showing red tissue color, no bleeding, collapsed to a depth of 2 - 4 mm from the buccal gingival margin; 3 = Socket filled with unorganized granulation tissue, more than ½ of the wound showing red tissue color, bleeding, no evidence of acute infection; 4 = Socket is filled with foreign material (food, etc.) and shows signs of alveolitis.

Changes in bone and soft tissue dimensions These will also be assessed on the same CBCT images taken at T0 (immediately postop) and T3 (4 months). Using specialized software (Invivo6, Osteoid Inc., Santa Clara, California, United States), both CBCT images are superimposed. The following reference lines will be constructed on the postoperative CBCT (T0) in the centre of the extracted tooth: the long axis of the extracted tooth, the level of the lingual bone crest perpendicular to the long axis of the extracted tooth, level -1 mm, level -3 mm and level -5 mm apical to the lingual bone crest and perpendicular to the long axis of the extracted tooth. Bone width is registered at the three levels -1, -3, and -5 mm. Buccal and lingual soft tissue height is measured as the vertical distance between the alveolar process and the soft tissue outline parallel to the vertical reference line at the most buccal and lingual part of the alveolar process. After completing all measurements on the postoperative CBCT, the software changes to the superimposed CBCT (T3) image so that the same measurements can be done while all keeping all reference lines. Finally, changes will be calculated by subtracting the measurements at T3 from the measurements at T0.

Changes in buccal soft tissue profile An intra-oral scan (Trios, 3shape, Copenhagen, Denmark) will be taken at T0 (immediately postop) and T3 (4 months). The obtained digital surface models in STL (Surface Tessellation Language) format will be imported into designated software (SMOP, Swissmeda AG, Zurich, Switzerland) to analyze profilometric changes. A study-relevant area of interest (AOI) at the buccal aspect is selected for each site. The AOI reaches from 0.5 mm below the soft tissue margin to 4 mm more apical. In mesiodistal dimension the AOI reaches from the mesial to the distal line angle. The AOI varies between sites due to individual anatomic differences but will be kept constant in each site across timepoints. Digital surface models are superimposed using the best-fit algorithm at the unchanged adjacent tooth surfaces. A mean volumetric change (mm3) within the AOI for each site from T0 to T3 is calculated by the software and divided by the AOI resulting in a mean change in buccal soft tissue profile. Details on the method can be found in an earlier paper (Eeckhout et al., 2020).

Statistical analysis SPSS Statistics 28 (IBM, New York, USA) will be used for data analysis. Mean values, standard deviations and 95% confidence intervals (CIs) will be calculated per treatment group. The paired samples t-test is used to compare test and control sites at 4 months in terms of soft tissue thickness in the centre of the site and buccal soft tissue profile.

A linear mixed model will be used to analyze the other secondary outcomes (horizontal buccal bone loss at the different levels, buccal and lingual soft tissue height, wound dimensions and SWHS). Treatment group, time, and their interaction will be modeled as fixed factors. Patient and tooth position as random factors. Estimated marginal means and 95% CIs will be calculated per treatment group and per timepoint. The level of significance is set at 0.05.

ELIGIBILITY:
Inclusion Criteria:

* At least 21 years old
* Good oral hygiene defined as a full-mouth plaque score ≤ 25% (O'Leary, Drake, & Naylor, 1972)
* Need for ARP after tooth extraction at two sites in the maxilla or mandible with > 50% buccal bone present following tooth extraction
* Signed informed consent

Exclusion Criteria:

* Any systemic disease
* Pregnancy
* Smoking (will be specifically asked)
* Untreated periodontitis
* Untreated caries lesions
* Suppuration and/or active infection around the failing tooth
* Midfacial recession at the failing tooth

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2024-01-02 (Actual); Primary Completion 2025-08-02 (Actual); Study Completion 2025-12-02 (Estimated)

PRIMARY OUTCOMES:
Soft tissue thickness in the centre of the site | pre-op, 4 months
  Changes in the soft tissue thickness at the centre of the site measured on CBCT

SECONDARY OUTCOMES:
Socket Wound Healing Score (SWHS) | 1 week, 3 weeks, 4 months
  SWHS is used to evaluate wound dehiscence, epithelialization, quality of granulation tissue filling the post-extraction socket, and depth between early granulation tissue and wound margin, score 0-4
Changes in bone and soft tissue dimensions | 4 months
  Changes in bone and soft tissue dimensions measured on CBCT images
Changes in buccal soft tissue profile | pre-op, 4 months
  Changes in buccal soft tissue profile measured by superimposing STL files using intra-oral scanners

CONTACTS AND LOCATIONS:
Locations (1):
- Ghent University Hospital, Ghent, East Flanders, Belgium

IPD SHARING:
Plan to Share IPD: Undecided
If the data can be included in a meta-analysis upon request by the authors, they can be transferred

REFERENCES:
- [Background] Afat IM, Akdogan ET, Gonul O. Effects of leukocyte- and platelet-rich fibrin alone and combined with hyaluronic acid on early soft tissue healing after surgical extraction of impacted mandibular third molars: A prospective clinical study. J Craniomaxillofac Surg. 2019 Feb;47(2):280-286. doi: 10.1016/j.jcms.2018.11.023. Epub 2018 Dec 3. PMID 30579747
- [Background] Avila-Ortiz G, Chambrone L, Vignoletti F. Effect of alveolar ridge preservation interventions following tooth extraction: A systematic review and meta-analysis. J Clin Periodontol. 2019 Jun;46 Suppl 21:195-223. doi: 10.1111/jcpe.13057. Erratum In: J Clin Periodontol. 2020 Jan;47(1):129. doi: 10.1111/jcpe.13212. PMID 30623987
- [Background] Eeckhout C, Bouckaert E, Verleyen D, De Bruyckere T, Cosyn J. A 3-Year Prospective Study on a Porcine-Derived Acellular Collagen Matrix to Re-Establish Convexity at the Buccal Aspect of Single Implants in the Molar Area: A Volumetric Analysis. J Clin Med. 2020 May 22;9(5):1568. doi: 10.3390/jcm9051568. PMID 32455863
- [Background] Martins JR, Wagner TP, Vallim AC, Konflanz W, Schwendicke F, Celeste RK, Haas AN. Comparison of the efficacy of different techniques to seal the alveolus during alveolar ridge preservation: Meta-regression and network meta-analysis. J Clin Periodontol. 2022 Jul;49(7):694-705. doi: 10.1111/jcpe.13628. Epub 2022 Apr 29. PMID 35451071
- [Background] O'Leary TJ, Drake RB, Naylor JE. The plaque control record. J Periodontol. 1972 Jan;43(1):38. doi: 10.1902/jop.1972.43.1.38. No abstract available. PMID 4500182
- [Background] Seyssens L, Eghbali A, Christiaens V, De Bruyckere T, Doornewaard R, Cosyn J. A one-year prospective study on alveolar ridge preservation using collagen-enriched deproteinized bovine bone mineral and saddle connective tissue graft: A cone beam computed tomography analysis. Clin Implant Dent Relat Res. 2019 Oct;21(5):853-861. doi: 10.1111/cid.12843. Epub 2019 Aug 28. PMID 31456345
- [Background] Tonetti MS, Cortellini P, Graziani F, Cairo F, Lang NP, Abundo R, Conforti GP, Marquardt S, Rasperini G, Silvestri M, Wallkamm B, Wetzel A. Immediate versus delayed implant placement after anterior single tooth extraction: the timing randomized controlled clinical trial. J Clin Periodontol. 2017 Feb;44(2):215-224. doi: 10.1111/jcpe.12666. Epub 2017 Jan 31. PMID 27978602